CLINICAL TRIAL: NCT04181554
Title: The Effect of Diastasis Recti on Postural Stability, Pelvic Floor Dysfunction and Respiratory Muscle Strength in Post-partum Women
Brief Title: Postural Stability, Pelvic Floor Dysfunction, Respiratory Muscle Strength in Post-partum Women With Diastasis Recti
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Hilal Denizoğlu Külli, Lecturer in Department of Physiotherapy and Rehabilitation, Bezmialem Vakif University
Other Study IDs: hdenizkulli3
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Diastasis Recti; Post-partum; Postural Stability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DRAM group: The post-partum women with DRAM
  Interventions: Other: Measurement of postural stability

INTERVENTIONS:
Other: Measurement of postural stability — The postural stability will assess by using Biodex balance system.

SUMMARY:
The aim of this study is to determine the effect of inter-rectus distance on postural stability, pelvic floor dysfunction and respiratory muscle strength in women with diastasis recti abdominis.

DETAILED DESCRIPTION:
Diastasis of recti abdominis muscles (DRAM) is defined as a separation of the two rectus abdominis muscles along the linea alba. Increased volume in the abdominal cavity, hormonal changes during pregnancy, neurodevelopmental differences, or abdominal wall laxity may caused. It is very common during pregnancy and may continue for eight weeks in postnatal period. The loss of abdominal wall stability and weakened pelvic floor muscles may occur with DRAM. The abdominal wall is one of the key point for body posture, trunk and pelvic stability. However, in our best knowledge, there is no study in the literature that evaluates women with and without DRA in terms of components related to postural control systems.

ELIGIBILITY:
Inclusion Criteria:

* Post- partum women (min 8 weeks - max 5 years)

Exclusion Criteria:

* Having a neurological, orthopedical or any other condition which affect postural stability.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The post-partum women with diastasis recti abdominis will be enrolled to the study.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Limits of stability test score | 5 minutes
  'Limits of Stability Test' will be performed using Biodex Balance System®. Subjects will stand on the platform and try to reach in eight directions spot that shown on the screen. The test results present scores for all eight directions and an overall score. Lower scores show worse performance (0= worst performance; 100= perfect performance)
Sensory integration test score | 6 minutes
  'Sensory integration test' will be performed using Biodex Balance System®. Volunteers will stand still on the platform in condition eyes open and closed on the firm and soft (foam) surfaces. The test scores are sway index for each condition and a composite score. Lower scores present better postural stability.

SECONDARY OUTCOMES:
Respiratory muscle strength | 5 minutes
  Inspiratory and expiratory muscle strength has been assessed by maximal inspiratory and expiratory mouth pressures.
Abdominal Muscle Endurance | 3 minutes
  Volunteers will be asked to perform curl up position as long as possible. The duration time will be measured until a maximum 180 seconds.
Pelvic floor dysfunction | 5 minutes
  Pelvic floor dysfunction will be assessed using "Pelvic Floor Distress Inventory". Lower scores show better pelvic floor functions.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Denizoglu Kulli, PhD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No